CLINICAL TRIAL: NCT01883128
Title: An Evaluation of a Novel Imaging Based Complex Diagnostic and Therapeutic Pathway Intervention for Men Who Fail Radiotherapy for Prostate Cancer.
Brief Title: FOcal RECurrent Assessment and Salvage Treatment
Acronym: FORECAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Hashim Uddin Ahmed, MRC Clinician Scientist and Clinical Lecturer in Urology, University College London Hospitals
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1R01CA135089 (NIH)
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Progression of Prostate Cancer
Keywords: Biochemical Failure; Radiotherapy; Radiorecurrent Prostate Cancer; MRI Prostate; Whole Body MRI; Bone Scan; Choline PET; Focal Salvage Treatment; HIFU; Cryotherapy

STUDY DESIGN:
Intervention Model Description: Whole-body MRI and Focal salvage therapy
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole body MRI (Experimental): Comparing the detection rate of metastases of whole body MRI compared to current standard of care tests - Choline PET and Bone scan.
  Interventions: Device: Whole Body MRI
- MRI Targeted Biopsies (Experimental): Transperineal MRI-targeted biopsies and whole-gland transperineal prostate mapping biopsies
  Interventions: Procedure: MRI Targeted biopsies
- Focal Salvage Therapy (Experimental): Focal salvage HIFU and cryotherapy of recurrent prostate cancer tumors only
  Interventions: Procedure: Focal Salvage Therapy

INTERVENTIONS:
Device: Whole Body MRI — Full parametric MRI using T1W, T2W, Diffusion-weighted and dynamic-contrast-enhanced images at 3Tesla
  Other Names: Philips Ingenia 3.0T Magnetic Resonance System; CE0344
  Arms: Whole body MRI
Procedure: Focal Salvage Therapy — Cryotherapy and HIFU will be used to targeted the areas of tumor only with a margin of normal tissue.
  Other Names: HIFU Device name: Sonablate 500; HIFU Device Serial Number 1049; Cryotherapy Device Name: Seed Net Gold; Cryotherapy Serial Number: Cat No FPRCH 2024
  Arms: Focal Salvage Therapy
Procedure: MRI Targeted biopsies — Image registration will be used to target biopsies followed by full mapping biopsies of the prostate. All biopsies will be carried out transperineally
  Other Names: SmartTarget software for image-registration
  Arms: MRI Targeted Biopsies

SUMMARY:
Radiotherapy is the commonest form of prostate cancer treatment in the UK. In one in four men, radiotherapy will fail to control the cancer. These men are offered hormonal treatment which has significant side effects. Few men are offered a further treatment such as surgery, HIFU or cryotherapy. Only half of these men are cancer free at 5 years. The investigators believe this is due to poor imaging tests such as CT and Bone scan that cannot accurately detect whether cancer has come back inside or outside of the prostate or both. Also radiotherapy damages tissue surrounding the prostate which affects tissue healing for example after surgery. Treating just the cancer in the prostate only (focal treatment) rather than the whole prostate may limit this damage and cause fewer side-effects. The investigators want to see if new imaging tests can better identify cancer that has spread outside of the prostate and areas of cancer inside the prostate. Our new tests are whole-body MRI (for distant disease) and MRI guided biopsies (MRI-TB) (for local disease). First, the investigators will compare the results of whole-body MRI to existing imaging tests (bone-scan, and choline PET/CT) that try to find distant spread. Second, the investigators will compare the results of MRI-TB to a very detailed and accurate biopsy of the prostate called template prostate mapping which will show us where and how aggressive the cancer is. Third, if the cancer is confined to the prostate, the investigators will treat men using focal salvage therapies HIFU and cryotherapy. The investigators believe that these new imaging tests could better identify those who will benefit from early hormone treatment and those who will benefit from local salvage treatment. Our study may help justify carrying out a larger trial looking at how good the treatment is in controlling cancer in the medium and long-term.

ELIGIBILITY:
Inclusion Criteria:

1. Previous external beam radiotherapy with or without neo-adjuvant/adjuvant hormone therapy
2. Biochemical failure as defined by the Phoenix criteria (PSA nadir + 2ng/ml)
3. Men considering local salvage treatment for radio-recurrent disease
4. Life expectancy of 5 years or more

Exclusion Criteria:

1. Have taken any form of hormones (except 5-alpha reductase inhibitors) within the previous 6 months
2. Unable to have MRI scan as defined by standard care practice
3. Metallic implant likely to cause artefact and reduce scan quality
4. PSA doubling time of 3 months or less
5. PSA value 20ng/ml or greater
6. Prior prostate biopsies following biochemical failure
7. Any prior local intervention to the prostate (e.g., laser/electrical resection or incision, cryotherapy, HIFU, any other ablative modality, any other radiotherapy, any other prostate injection therapy for symptoms or cancer control)
8. Unable to have general or regional anaesthesia
9. Unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of whole body MRI in identifying distant disease | 2 years
  Whole body MRI lesions suspicious of lymph node, visceral or bone metastases compared to standard care tests
  - Sensitivity, specificity, negative and positive predictive values of whole-body MRI to detect distant disease compared to standard care tests (isotope bone-scan, PET/CT-scan, with skeletal survey where appropriate) and/or pelvic lymphadenectomy and/or biopsy of distant areas in indeterminate cases

SECONDARY OUTCOMES:
Can multiparametric MRI accurately detect localised recurrent prostate cancer | 2 years
  Imaging of Local Disease
  Transperineal multi-parametric MRI targeted biopsies compared to Template Prostate Mapping biopsies in the detection of UCL definition 2 clinically significant prostate cancer (Gleason >/=3+4 AND/OR Maximum Cancer Core Length >/=4mm in any one biopsy)

OTHER OUTCOMES:
To determine urinary incontinence rates after focal salvage therapy to localised recurrent prostate cancer? | 2 years
  Treatment
  Continence Presence of urinary incontinence (any pad usage) as determined by the UCLA-EPIC urinary continence questionnaire, at 12 months, in those men with no urinary incontinence at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, FRCS, PhD, Study Chair — University College London Hospitals; Manit Arya, FRCS, Principal Investigator — University College London Hospitals; Mark Emberton, FRCS, MD, Principal Investigator — University College London Hospitals; Shonit Punwani, FRCR, Principal Investigator — University College London Hospitals
Locations (2):
- United Kingdom (2):
  - Hampshire Hospitals NHS Trust, London
  - University College London Hospitals, London

REFERENCES:
- [Derived] Light A, Kanthabalan A, Otieno M, Pavlou M, Omar R, Adeleke S, Giganti F, Brew-Graves C, Williams NR, Emara A, Haroon A, Latifoltojar A, Sidhu H, Freeman A, Orczyk C, Nikapota A, Dudderidge T, Hindley RG, Virdi J, Arya M, Payne H, Mitra AV, Bomanji J, Winkler M, Horan G, Moore CM, Emberton M, Punwani S, Ahmed HU, Shah TT. The Role of Multiparametric MRI and MRI-targeted Biopsy in the Diagnosis of Radiorecurrent Prostate Cancer: An Analysis from the FORECAST Trial. Eur Urol. 2024 Jan;85(1):35-46. doi: 10.1016/j.eururo.2023.09.001. Epub 2023 Sep 29. PMID 37778954
- [Derived] Light A, Peters M, Reddy D, Kanthabalan A, Otieno M, Pavlou M, Omar R, Adeleke S, Giganti F, Brew-Graves C, Williams NR, Emara A, Haroon A, Latifoltojar A, Sidhu H, Freeman A, Orczyk C, Nikapota A, Dudderidge T, Hindley RG, Virdi J, Arya M, Payne H, Mitra AV, Bomanji J, Winkler M, Horan G, Moore C, Emberton M, Punwani S, Ahmed HU, Shah TT. External validation of a risk model predicting failure of salvage focal ablation for prostate cancer. BJU Int. 2023 Nov;132(5):520-530. doi: 10.1111/bju.16102. Epub 2023 Jun 29. PMID 37385981
- [Derived] Shah TT, Kanthabalan A, Otieno M, Pavlou M, Omar R, Adeleke S, Giganti F, Brew-Graves C, Williams NR, Grierson J, Miah H, Emara A, Haroon A, Latifoltojar A, Sidhu H, Clemente J, Freeman A, Orczyk C, Nikapota A, Dudderidge T, Hindley RG, Virdi J, Arya M, Payne H, Mitra A, Bomanji J, Winkler M, Horan G, Moore CM, Emberton M, Punwani S, Ahmed HU. Magnetic Resonance Imaging and Targeted Biopsies Compared to Transperineal Mapping Biopsies Before Focal Ablation in Localised and Metastatic Recurrent Prostate Cancer After Radiotherapy. Eur Urol. 2022 Jun;81(6):598-605. doi: 10.1016/j.eururo.2022.02.022. Epub 2022 Mar 31. PMID 35370021